CLINICAL TRIAL: NCT05863442
Title: A First-in-human, Randomized, Double-blind, Parallel-group Study to Evaluate the PK, Safety, Tolerability, Immunogenicity, and PD Profile of a Single Intravenous Dose of TUR03 Compared With Soliris® in Healthy Adult Male Participants
Brief Title: Comparative PK, Safety, Tolerability, Immunogenicity, and PD Profile Study of TUR03 and Soliris in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turgut Ardika PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TUR03-22-01
Record Dates: First submitted 2023-03-17; First posted 2023-05-18 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: eculizumab; phase I; biosimilar
MeSH Terms: interventions — eculizumab; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soliris (Active Comparator)
  Interventions: Drug: Soliris 300 MG in 30 ML Injection
- TUR03 (Experimental)
  Interventions: Drug: TUR03 300 MG in 30 ML Injection

INTERVENTIONS:
Drug: Soliris 300 MG in 30 ML Injection — Active Comparator
  Arms: Soliris
Drug: TUR03 300 MG in 30 ML Injection — Investigational medicinal Product, eculizumab - Turgut
  Arms: TUR03

SUMMARY:
This study is designed as a randomized, double-blind, parallel-group study to evaluate the PK, safety, tolerability, immunogenicity, and PD of TUR03 compared to Soliris, when administered as a single IV infusion in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if ALL of the following criteria apply:

1. Capable of giving signed informed consent as described in Section 10.1, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol.
2. Participants assigned male at birth who are ≥18 years and ≤45 years old at the time of signing the ICF.
3. Body weight ≥50 kg and ≤90 kg and body mass index (BMI) ≥18.00 kg/m2 and ≤30.00 kg/m2 at Screening and Day -1.
4. Participants must be healthy as determined by the Investigator, based on medical history, physical examination, vital signs, ECG, and clinical laboratory evaluations at Screening and Day -1, as follows:

   1. Hematology and coagulation results within reference ranges.
   2. Liver function panel analyte values ≤1.5 × upper limits of normal (ULN), which include aspartate transaminase, alanine transaminase, and total bilirubin (for participants with Gilbert's Syndrome, total bilirubin ≤3.0 × ULN is allowed if direct bilirubin is ≤50%), alkaline phosphatase, and gamma glutamyl transferase at Screening.
   3. Urinalysis within reference ranges or showing no clinically significant findings.

   NOTE: One repeat of clinical laboratory tests is allowed at the discretion of the Investigator.
5. Participants must have documented evidence of prior complete vaccination with meningococcal vaccines against N. meningitidis serogroup B at any time and against serogroups A, C, W, and Y within 5 years prior to Screening in line with local immunization requirements or must agree to be vaccinated against N. meningitidis during the study.
6. Nonsterilized participants with partners of childbearing potential must agree to take appropriate contraceptive measures (as described in Section 10.4) from Day 1 until 5 months after IP administration and refrain from donating sperm during this period. NOTE: Participants with pregnant partners are excluded.
7. Nonsmoker or occasional smoker, ie, smokes ≤10 cigarettes (or equivalent of tobacco- or nicotine-containing products) per week within 30 days prior to Screening and is able to abide by the smoking policy of the study site.
8. Ability and willingness to abstain from alcohol from 48 hours before admission to the study site on Day -1, during in-house observation at the study site until discharge, and for 24 hours prior to ambulatory visits.

Exclusion Criteria:

Participants are excluded from the study if ANY of the following criteria apply:

1. Known or suspected hereditary or acquired complement deficiency.
2. History of meningococcal infection.
3. History or evidence of a clinically significant disorder (including psychiatric disorders), condition, or disease that, in the opinion of the Investigator and Medical Monitor or designee, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion. EXCEPTION: Fully resolved childhood asthma is not exclusionary.
4. History of splenectomy.
5. History of surgery or major trauma within 12 weeks of Screening, or surgery planned during the study.
6. A recent history (within 1 week prior to IP administration) or presence or suspicion of current active systemic or local infection, a known risk for developing sepsis, and/or known active inflammatory condition, in the opinion of the Investigator.
7. History of or current invasive malignancy (excluding basal or squamous cell carcinoma that has been fully resected with no evidence of metastatic disease for 1 year).
8. History of ongoing seborrheic dermatitis or eczema.
9. History of clinically significant headaches that, in the opinion of the Investigator, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
10. History of recurrent/chronic hemorrhages or any hemorrhage within 30 days prior to IP administration.
11. History of a drug- or food-induced severe hypersensitivity reaction (eg, immunologic or nonimmunologic anaphylaxis).
12. Known hypersensitivity reaction to penicillin and/or cephalosporin that, in the opinion of the Investigator, would pose a risk to participant safety.
13. Known hypersensitivity to any component of TUR03 or Soliris, murine proteins, or other monoclonal antibodies.
14. Known hypersensitivity to any component of meningococcal vaccines, including those containing diphtheria toxoid, or a life-threatening reaction after previous administration of a vaccine containing similar components.
15. Hypertension at Screening or Day -1 (defined as a systolic blood pressure [BP] >140 mm Hg and/or a diastolic BP >90 mm Hg, confirmed by a single repeat measurement that same day) or a history of hypertension requiring pharmacological intervention.
16. Proteinuria at Screening or Day -1 (with a urine dipstick value of 1+ or above)..
17. Tests positive for human immunodeficiency virus (HIV 1 and 2), hepatitis B virus surface antigen, hepatitis B core antibody, or hepatitis C virus.
18. Tests positive for tuberculosis (TB) using the QuantiFERON®-TB Gold test at Screening or, if indeterminant result on the first test, tests positive or indeterminant on repeat QuantiFERON-TB Gold test.
19. Positive screen for alcohol by breath test and/or potential drugs of abuse by urine drug screen at Screening or Day -1. NOTE: One repeat screen is allowed at the discretion of the Investigator.
20. History of alcohol or drug abuse or drug addiction (including cannabis products) within the last 12 months prior to Screening.
21. Prior exposure to eculizumab or similar compounds (ie, a monoclonal antibody that specifically binds to the complement protein C5).
22. Use of immunoglobulins or iron supplementation within 3 months prior to Screening.
23. Use of any over-the-counter (OTC) medications, herbal remedies such as St. John's Wort extract, or prescription medications within 7 days or 5 half lives (whichever is longer) prior to IP administration. EXCEPTIONS: Vitamins, dietary supplements, and paracetamol (up to 4 g per day, but <1 g in 4 hours) for analgesia are not exclusionary.
24. Use of other investigational drugs (or is currently using an investigational device) within 60 days or 5 half-lives (whichever is longer) prior to IP administration.
25. Vaccination with a live vaccine within 30 days prior to IP administration, or vaccination with an inactivated vaccine or approved COVID-19 vaccine within 14 days prior to IP administration, or planning to get vaccinated during the study period. EXCEPTIONS: Receipt of required meningococcal vaccinations per protocol is not exclusionary.
26. Veins unsuitable for venous blood collection.
27. Donated blood (including blood products) or experienced loss of blood ≥500 mL within 30 days of Screening, or donated plasma within 7 days of Screening.
28. Participant is a family member or employee of the Investigator or Sponsor.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-07-23 (Estimated); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
PK similarity of TUR03 and Soliris following a single IV infusion in healthy participants | Day 1 - Day 57
  The primary endpoint for PK similarity is AUC(0-inf).

SECONDARY OUTCOMES:
Eculizumab serum concentration-time profile | Day 1 - Day 57
  Serum eculizumab concentrations will be listed and summarized using descriptive statistics by treatment group and nominal PK sampling time point. All serum eculizumab concentrations that are below the limit of quantification will be labeled as such in the concentration data listings. Individual and arithmetic mean (per treatment) concentration-time profiles will also be presented graphically.
Maximum serum concentration (Cmax) | Day 1- Day 57
  Observed concentration versus time data
Area under the concentration-time curve from time zero to the last quantifiable concentration (AUClast) | Day 1- Day 57
  AUC(0-last)
Time to Cmax | Day 1 - Day 57
  tmax
Terminal half-life | Day 1 - Day 57
  t½
Volume of distribution during terminal phase after intravenous administration | Day 1 - Day 57
  Vz
Terminal elimination rate constant | Day 1 - Day 57
  Kel
Total serum clearance of drug after intravenous administration | Day 1 - Day 57
  CL
AEs and AESI | Day 1 - Day 57
  infusion-related reactions, meningococcal infections, and other serious systemic infections
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Hematology | Day 1 - Day 57
  Platelet count, Red blood cell count, Neutrophils, Hemoglobin, Lymphocytes, Hematocrit, Monocytes, Eosinophils, Mean corpuscular volume, Basophils, Mean corpuscular hemoglobin, Mean cell hemoglobin concentration will be measured to assess changes in hematological parameters in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Coagulation - International normalized ratio | Day 1 - Day 57
  International normalized ratio (INR) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Coagulation - Activated partial thromboplastin time | Day 1 - Day 57
  Activated partial thromboplastin time (sec) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Coagulation - Prothrombin time | Day 1 - Day 57
  Prothrombin time (sec) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Urea | Day 1 - Day 57
  Urea (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Carbon dioxide (bicarbonate) | Day 1 - Day 57
  Carbon dioxide (bicarbonate)(mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Creatinine | Day 1 - Day 57
  Creatinine (mcmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - AST | Day 1 - Day 57
  AST (U/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - ALT | Day 1 - Day 57
  ALT (U/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - ALP | Day 1 - Day 57
  ALP (U/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Glucose (fasting) | Day 1 - Day 57
  Glucose (fasting)(mcmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Gamma glutamyl transferase | Day 1 - Day 57
  Gamma glutamyl transferase (U/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Total Protein | Day 1 - Day 57
  Total protein (g/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Creatine kinase | Day 1 - Day 57
  Creatine kinase (U/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Potassium | Day 1 - Day 57
  Potassium (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Lactate dehydrogenase | Day 1 - Day 57
  Lactate dehydrogenase (U/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Sodium | Day 1 - Day 57
  Sodium (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Albumin | Day 1 - Day 57
  Albumin (g/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Chloride | Day 1 - Day 57
  Chloride (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Total and direct bilirubin | Day 1 - Day 57
  Total and direct bilirubin (mcmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Calcium | Day 1 - Day 57
  Calcium (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Triglycerides | Day 1 - Day 57
  Triglycerides (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Phosphate | Day 1 - Day 57
  Phosphate (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Clinical chemistry - Cholesterol | Day 1 - Day 57
  Cholesterol (mmol/L) will be measured in blood samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Leukocytes | Day 1 - Day 57
  Leukocytes, will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Red blood cells | Day 1 - Day 57
  Red blood cells (/hpf) will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Protein | Day 1 - Day 57
  Protein (mg/dL) will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - pH | Day 1 - Day 57
  pH will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Bilirubin | Day 1 - Day 57
  Bilirubin will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Nitrite | Day 1 - Day 57
  Nitrite will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Urobilinogen | Day 1 - Day 57
  Urobilinogen (EU/dl) will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Specific gravity | Day 1 - Day 57
  Specific gravity will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Ketones | Day 1 - Day 57
  Ketones (mg/dL) will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Glucose | Day 1 - Day 57
  Glucose (mg/dL) will be measured to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Incidence of Treatment-Emergent changes in safety clinical laboratory parameters from baseline and Grade 3 laboratory abnormalities - Urinanalysis - Microscopy | Day 1 - Day 57
  Microscopic (if clinically indicated)(/hpf) analyses to assess changes in urine-related parameters in urine samples. Any clinically significant pathology results (that require reporting as an adverse event) will be incorporated into the adverse event table.
Changes in vital signs - Blood Pressure | Day 1 - Day 57
  Systolic and diastolic blood pressure will be assessed with a completely automated device. Wherever possible, vital signs measurements must be taken using the same body position at subsequent visits and consistent methods between participants.
Changes in vital signs - Pulse rate | Day 1 - Day 57
  Pulse rate will be assessed with a completely automated device. Wherever possible, vital signs measurements must be taken using the same body position at subsequent visits and consistent methods between participants.
Changes in vital signs - Body Temperature | Day 1 - Day 57
  Body temperature (aural is preferred), will be assessed with a completely automated device. Wherever possible, vital signs measurements must be taken using the same body position at subsequent visits and consistent methods between participants.
Changes in Electrocardiograms (ECG) - Heart rate | Day 1 - Day 57
  Single 12-lead ECGs will be obtained after the participant has rested comfortably in the supine position for at least 5 minutes in a quiet setting without distractions (eg, television, cell phones) using an ECG machine that automatically calculates the heart rate. All ECG data will be documented at each prespecified time point, and the details will be recorded in both the source documents and the eCRF. The Investigator (or a qualified delegate at the investigational site) will interpret the ECG using 1 of the following categories: normal, abnormal not clinically significant, or abnormal clinically significant and record their evaluation in the eCRF.
Changes in Electrocardiograms (ECG) - PR interval | Day 1 - Day 57
  Single 12-lead ECGs will be obtained after the participant has rested comfortably in the supine position for at least 5 minutes in a quiet setting without distractions (eg, television, cell phones) using an ECG machine that automatically measures PR interval. All ECG data will be documented at each prespecified time point, and the details will be recorded in both the source documents and the eCRF. The Investigator (or a qualified delegate at the investigational site) will interpret the ECG using 1 of the following categories: normal, abnormal not clinically significant, or abnormal clinically significant and record their evaluation in the eCRF.
Changes in Electrocardiograms (ECG) - RR interval | Day 1 - Day 57
  Single 12-lead ECGs will be obtained after the participant has rested comfortably in the supine position for at least 5 minutes in a quiet setting without distractions (eg, television, cell phones) using an ECG machine that automatically measures RR interval. All ECG data will be documented at each prespecified time point, and the details will be recorded in both the source documents and the eCRF. The Investigator (or a qualified delegate at the investigational site) will interpret the ECG using 1 of the following categories: normal, abnormal not clinically significant, or abnormal clinically significant and record their evaluation in the eCRF.
Changes in Electrocardiograms (ECG) - QRS duration | Day 1 - Day 57
  Single 12-lead ECGs will be obtained after the participant has rested comfortably in the supine position for at least 5 minutes in a quiet setting without distractions (eg, television, cell phones) using an ECG machine that automatically measures QRS duration. All ECG data will be documented at each prespecified time point, and the details will be recorded in both the source documents and the eCRF. The Investigator (or a qualified delegate at the investigational site) will interpret the ECG using 1 of the following categories: normal, abnormal not clinically significant, or abnormal clinically significant and record their evaluation in the eCRF.
Changes in Electrocardiograms (ECG) - QT interval | Day 1 - Day 57
  Single 12-lead ECGs will be obtained after the participant has rested comfortably in the supine position for at least 5 minutes in a quiet setting without distractions (eg, television, cell phones) using an ECG machine that automatically measures QT interval. The QT interval corrected for heart rate by Fridericia's formula (QTcF interval) will be derived. All ECG data will be documented at each prespecified time point, and the details will be recorded in both the source documents and the eCRF. The Investigator (or a qualified delegate at the investigational site) will interpret the ECG using 1 of the following categories: normal, abnormal not clinically significant, or abnormal clinically significant and record their evaluation in the eCRF.
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 via physical examination | Day 1 - Day 57
  Complete physical examination will be performed by a study-delegated registered physician at Screening and will include, at a minimum, assessments of general appearance, head, ears, eyes, nose, throat, neck (including thyroid), skin, cardiovascular system, respiratory, system, gastrointestinal system, musculoskeletal system, lymph nodes, and nervous system. A brief physical examination will be performed at specified time points outlined in the SoA and will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). A symptom-directed physical examination, including areas with previously noted abnormalities and/or that are associated with any new complaints from the participant, will be performed at all other visits and at any time throughout the study, as clinically indicated.
Comparison of the immunogenicity of TUR03 and Soliris following a single IV infusion in healthy participants - Frequency of antidrug antibodies (ADAs) | Day 1 - Day 57
  Frequency of ADAs will be assessed. Serum samples will be screened for antibodies binding to eculizumab in TUR03 and Soliris. The detection and characterization of ADAs to eculizumab will be performed using validated immunoassay methods.
Comparison of the immunogenicity of TUR03 and Soliris following a single IV infusion in healthy participants - Antidrug antibody titers | Day 1 - Day 57
  Titers of ADAs will be assessed.
Comparison of the immunogenicity of TUR03 and Soliris following a single IV infusion in healthy participants - Neutralizing antibodies (NAbs) | Day 1 - Day 57
  The frequency of NAbs will be assessed in ADA-positive participants' sera. Subsequent to the confirmation of ADA-positivity, antibodies will be further characterized and evaluated for their ability to neutralize the activity of the IP (TUR03 and Soliris).
PD profile of TUR03 and Soliris - ABEC (0-1344) CH50 | Day 1 - Day 57
  Area between the baseline and effect curves for hemolytic complement activity from 0 to 1344 hours
PD profile of TUR03 and Soliris - AUEC(0-1344) CH50 | Day 1 - Day 57
  Area under the effect curve for hemolytic complement activity from 0 to 1344 hours
PD profile of TUR03 and Soliris - Emin CH50 | Day 1 - Day 57
  Minimum hemolytic complement activity from 0 to 1344 hours
PD profile of TUR03 and Soliris - Tmin CH50 | Day 1 - Day 57
  Time to minimum hemolytic complement activity from 0 to 1344 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Limited, Herston, Queensland, Australia